CLINICAL TRIAL: NCT05623306
Title: A Double-Blinded, Randomized, Crossover Trial of Stereoencephalography- Guided Multi-Lead Deep Brain Stimulation for Treatment-Refractory Obsessive- Compulsive Disorder (SEEG-Guided DBS for OCD)
Brief Title: SEEG-Guided DBS for OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Casey H. Halpern, M.D. (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Casey H. Halpern, M.D., Associate Professor of Neurosurgery, Director of Stereotactic and Functional Neurosurgery, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 851810
Record Dates: First submitted 2022-10-14; First posted 2022-11-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Stage 1: Invasive SEEG Monitoring and Recovery
  Stage 2: SEEG-guided DBS Implantation and Optimization of DBS Programming
  Stage 3: Randomized Sham-controlled Crossover Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SEEG Guided DBS ON-OFF (Stimulation-Sham) (Experimental): Patients in the ON-OFF arm will first be treated for up to 12 weeks with the parameters identified during the DBS optimization phase until the washout period.
  Interventions: Device: PMT Stereoencephalography (SEEG); Device: Vercise Genus™ Deep Brain Stimulation (DBS) System or Percept™ PC Neurostimulation System
- SEEG Guided DBS OFF-ON (Sham-Stimulation) (Sham Comparator): Patients in the OFF-ON will have their devices turned off and will not have their device switched on (activated) until the crossover point.
  Interventions: Device: PMT Stereoencephalography (SEEG); Device: Vercise Genus™ Deep Brain Stimulation (DBS) System or Percept™ PC Neurostimulation System

INTERVENTIONS:
Device: PMT Stereoencephalography (SEEG) — For Stage 1 of this study, we will be implanting depth electrodes to record stereoencephalography across a network of brain regions.
  Other Names: Ad-Tech Depth Electrodes
Device: Vercise Genus™ Deep Brain Stimulation (DBS) System or Percept™ PC Neurostimulation System — For Stages 2 and 3 of this study, we intend to use the DBS system to treat patients with severe symptoms of chronic, treatment-refractory OCD by targeting stimulation to sites that have been determined to have therapeutic benefit during our SEEG Invasive Monitoring phase.

SUMMARY:
This is a multi-site, double-blinded, randomized, crossover study design for SEEG-guided 4-lead DBS for treatment-refractory OCD, followed by open label stimulation for an additional 6 months. The study will be conducted in 3 stages: Stage 1 will consist of SEEG brain mapping and optimization of stimulation parameters. Stage 2 will consist of DBS surgery and further optimization of stimulation parameters. Stage 3 will be randomized, crossover treatment, followed by open label treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 22 years and ≤ 75 years of age, at the time of screening
2. Chronic (> 5 years preceding the date of enrollment) OCD, diagnosed as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition guidelines (DSM-5)

   1. Presence of obsessions, compulsions, or both
   2. Time-consuming obsessions and compulsions that take more than one hour a day or cause clinically significant distress or impairment in social, occupational, or other important areas of functioning
   3. Obsessive-compulsive symptoms that are not attributable to the physiological effects of a substance (e.g. a drug of abuse, a medication) or another medical condition
   4. Disturbance not better explained by the symptoms of another mental disorder listed in the DSM-5
3. Severe OCD symptoms, as defined by Y-BOCS I score of ≥ 28, within two weeks prior to enrollment
4. Lack of adequate response to a history of the following treatments, based on information from any of the following: (a) the current treating physician and/or psychologist; (b) medical records or other forms of communication from previous healthcare providers; and (c) pharmacy records, as determined by the Principal Investigator

   1. Adequate trial of ≥ 2 selective serotonin reuptake inhibitors (SSRIs) for an adequate duration at the maximum dose recommended for OCD or at the maximally-tolerated dose according to the FDA-approved package labeling
   2. Adequate trial of ≥ 1 augmentation trial using an antipsychotic medication
   3. Adequate trial of clomipramine, either as monotherapy or as an augmentation therapy, unless medically contradicted
   4. Adequate trials of cognitive behavior therapy-based Exposure and Response Prevention (ERP)
5. Willingness and ability to remain on the same daily dose of any and all scheduled psychotropic medication(s) for at least 8 weeks prior to study enrollment and for the duration of the trial, as determined by the research/study psychiatrist and the PI
6. Willingness and ability to discontinue any psychotherapeutic behavioral intervention therapy (e.g. CBT) until the maintenance stage, if any, as determined safe by the research/study psychiatrist
7. Study participation in the prospective subject's best psychiatric interest, as determined by the research/study psychiatrist and based on a comprehensive assessment that includes the following: (a) detailed psychiatric history; (b) examination of the mental status; (c) review of psychiatric assessment measures obtained to determine eligibility, as applicable; (d) review of previous medical records for a minimum of 2 years prior to enrollment, or as applicable; and (e) consideration of the potential benefits versus risks of study participation
8. Agreement to being evaluated by a licensed psychiatrist and/or psychologist at regular intervals, as required by the schedule of events, for the duration of study participation
9. Living within 6 hours of driving distance from study sites and no plan of relocation for at least the duration of the trial (approximately 18-24 months), as reported by the prospective subject or a family member
10. Adequate social support, including but not limited to, stable housing and two family members and/or friends, who are identified as a verifiable emergency contacts
11. Willingness and ability to provide at least two verifiable contacts for emergency purposes and to permit verification of emergency contacts by research staff before all study visits and as needed, at the discretion of the Principal Investigator
12. Ability to understand procedure-related instructions and to complete study assessments in English, in the opinion of the Principal Investigator
13. Willingness and ability to comply with protocol requirements (e.g. procedure visits, treatment schedule, follow-up visit schedule, evaluations, etc.), in the opinion of the Principal Investigator
14. Willingness and ability to provide written agreement to allow any and all forms of communication between the research team and treating clinician(s)
15. Willingness and ability to provide informed consent, in the opinion of the Principal Investigator

Exclusion Criteria:

1. Diagnosis of, according to the Mini International Neuropsychiatric Interview (MINI), any other primary psychiatric diagnosis defined in the DSM-5, including Hoarding Disorder.

   a. Subjects with secondary psychiatric diagnosis will not be excluded, except as described below.
2. In the opinion of the Principal Investigator and relative to the date of enrollment, (a) current or past diagnosis of, or medical history/records suggestive of, a DSM-5 defined Personality Disorder, considered to be severe; or (b) history of hospitalization because of Borderline Personality Disorder
3. Clinical secondary diagnosis made by a psychiatrist, as defined in the DSM-5 and based on the MINI and the psychiatric evaluation:

   1. Lifetime diagnosis of Bipolar I Disorder or Bipolar II Disorder
   2. Current/active diagnosis of Anorexia Nervosa, Bulimia Nervosa, or Binge Eating Disorder

   i. Diagnosis will be considered current/active if the subject had an active episode within 5 years of screening. c. Lifetime diagnosis of a primary psychotic disorder (e.g. Schizophrenia, Schizoaffective Disorder) d. Current/active diagnosis of mood disorder with psychotic features i. Diagnosis will be considered current/active if the subject had an active episode within 2 years of screening.
4. Current suicidal risk, as determined by the research/study psychiatrist using the brief mental status exam and the psychiatric interview (including the Columbia Suicide Severity Rating Scale [C-SSRS]), or significant suicide risk, defined as Hamilton Depression Rating Scale (HDRS-21) Item 3 score of ≥ 3 or any lifetime history of suicide attempt

   a. Subjects who answer 'Yes' to questions 3, 4, or 5 of the C-SSRS will be excluded.
5. Treatment, within two years of screening, for any of the following: dependency on, addiction to, use of, abuse of, or overuse of any illicit substance(s), including alcohol, but not including nicotine or caffeine
6. History of head trauma associated with any of the following:

   1. Loss of consciousness for > 5 minutes
   2. A residual effect(s) that failed to resolve completely at least 1 year prior to the date of screening
   3. An abnormality on a neuroimaging study (MRI, CT Scan) that was/is attributable to the head trauma
   4. > 1 head injury within the past 2 years which were diagnosed as a concussion, concussive-type or traumatic brain injury (TBI), according to medical records or as reported by the prospective subject or a family member
7. Any of the following permanent implants:

   1. Cardiac implant (e.g. pacemaker or any intracardiac lines, implanted neurostimulators, shunts)
   2. Brain implant (e.g. intracranial implant, aneurysm clips, shunts, stimulators, cochlear implants, or electrodes)
   3. Implanted medical pumps
8. Diathermy treatments requirement for any reason
9. Hearing loss that, in the opinion of the Principal Investigator, an audiologist, or a treating physician, is likely to affect the subject's ability to comply with all of the requirements of the study or may affect the integrity of the study data
10. Any metal or metallic particles anywhere in the head, except in the inside of the mouth
11. Pregnancy, at the time of screening or during the course of the study (i.e. 3 years)

    a. Acceptable methods of contraception include the following: i. Established use of oral, injected or implanted contraceptives ii. Placement of an intrauterine device (IUD) or an intrauterine system (IUS) iii. Female sterilization (e.g. surgical bilateral oophorectomy with or without hysterectomy, total hysterectomy, tubal ligation) iv. Male sterilization, with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate v. True abstinence, when in line with the preferred and usual lifestyle of the subject b. Barrier methods of contraception, such as a condom, a diaphragm, or cervical/vault caps with spermicidal foam/gel/film/cream/suppository, and rhythm methods of contraception, although encouraged, alone are not considered acceptable forms or contraception.
12. History of involuntary movements, in the opinion of the Principal Investigator or a neuro-radiologist
13. History of excessive or prolonged bleeding and/or any of the following:

    1. INR of > 1.8
    2. Prolonged activated partial thromboplastin time (aPTT) of ≥ 45 sec
    3. Platelet count of < 100×100/L
14. Allergy to gadolinium
15. Inability to safely and successfully undergo an MRI or a CT Scan
16. Any past or present medical condition, disease, disorder, or injury that, in the opinion of the Principal Investigator, may reduce or hinder the subject's ability to fully comply with all study requirements for the duration of the study or may impact, compromise, or affect the integrity of the data or the results of the study
17. Current participation in other research that may potentially interfere with DBS study objectives or with the ability to follow the timeline of this study, as determined by the Principal Investigator

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Endpoint #1 - OCD Relevant Network | 14 days
  Percentage of patients in which an OCD relevant network can be identified
Primary Feasibility Endpoint #2 - Stimulation Target That Acutely Improves OCD Symptoms | 14 days
  Percentage of patients in which we can identify a stimulation target that acutely improves OCD symptoms during SEEG Stage 1
Primary Feasibility Endpoint #3 - Willingness to Continue with DBS Stage 2 | Day 14
  Percentage of patients willing and able to continue with the DBS Stage 2 after completing the SEEG Stage 1
Primary Feasibility Endpoint #4 - Acute Symptomatic Improvement | Approximately 60 weeks
  Percentage of implanted DBS sites associated with both acute symptomatic improvement during the SEEG Stage 1 and therapeutic benefit during the DBS Stage 2.
Primary Efficacy Endpoint - Treatment Response | Up to 24 weeks
  Treatment response, determined by the difference in Y-BOCS II score between the active stimulation (ON) condition and sham control (OFF) condition
Primary Safety Endpoint - Serious Adverse Events | Approximately 4 years
  Number and type of serious adverse events in this SEEG-guided 4-lead DBS approach compared to conventional DBS for OCD.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP